CLINICAL TRIAL: NCT02586168
Title: The Effect of Gemcabene (CI-1027) on Insulin Sensitivity in Nondiabetic Subjects
Brief Title: The Effect of Gemcabene on Insulin Sensitivity in Nondiabetic Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NeuroBo Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 1027-014
Record Dates: First submitted 2015-10-22; First posted 2015-10-26 (Estimated); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Insulin Sensitivity
Keywords: Insulin Resistance; Lipid Regulator
MeSH Terms: conditions — Insulin Resistance | interventions — gemcabene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gemcabene 900 mg (Experimental): Gemcabene 900 mg
  Interventions: Drug: Gemcabene 900 mg
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gemcabene 900 mg — Gemcabene 900 mg once daily (QD)
  Arms: Gemcabene 900 mg
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effect of gemcabene on insulin sensitivity as defined by average glucose disposal rate.

ELIGIBILITY:
Inclusion Criteria:

* Good health, as determined by medical history, physical examination, EKG and clinical laboratory assessments
* Males; and females of non-reproductive potential
* Obesity
* Non-diabetic

Exclusion Criteria:

* Use of any medication considered unacceptable by the clinical investigators during the 14-day period before the start of Day 1. Hormone Replacement Therapy is acceptable.
* Use of a lipid-lowering agent (niacin, fibrates, statin) during the 8 weeks before screening
* Use of any anti-diabetic medications
* Use of any steroid medications
* Donation of any blood or plasma product or participation in another study in the 30 days prior to Day 1
* If female, pregnant, lactating or of childbearing potential; and
* History of significant reaction to any fibrate lipid-lowering agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2001-07; Primary Completion 2001-10 (Actual); Study Completion 2001-10 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | 4 weeks

SECONDARY OUTCOMES:
Adverse Events | 4 weeks
ECG | 4 weeks
  Clinically Significant Changes
Clinical Laboratory - hematology, chemistry | 4 weeks
  Clinical Laboratory Abnormalities